CLINICAL TRIAL: NCT06593808
Title: SOon HOme Study. Early Open Cot Transfer in Preterm Infants, a Randomized Controlled Trial
Brief Title: SOon HOme Study About Preterm Infants
Acronym: SOHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6575
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preterm Birth Complication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm infants in incubator (No Intervention): Preterm infant in stable conditions transferred from the incubator to the open crib at a weight greater than or equal to 1600 grams
- Preterm infants in open coat (Experimental): Preterm infant in stable conditions transferred from the incubator to the open crib at a weight greater than or equal to 1400 grams
  Interventions: Procedure: Weaning from the incubator to open coat at a weight greater than or equal to 1400 grams

INTERVENTIONS:
Procedure: Weaning from the incubator to open coat at a weight greater than or equal to 1400 grams — They will be dressed in a woolen hat and dress, wrapped in a blanket and placed in crib with preheated mattress.Vital signs will be monitored daily.Axillary temperature will be measured every 3 hours for the first 12 hours, if above or equal to 36.5°C it will be measured every 6 hours for the next 36 hours. If normothermia for 48 hours, the preheated mattress will be turned off and temperature monitoring will be continued every 3 hours for 24 hours.If greater than or equal to 36.5°C, thermal control will be continued every 8 hours for 48 hours, at the end of which time, if normothermic, care will be confirmed.If not it will be placed back in the crib with heated mattress.If temperature still below 36.5°C, an additional blanket will be placed and it will be rechecked after 2 hours.If it remains below 36.5°C, the infant will be placed under a radiant lamp and the temperature will be checked after 3 hours.If hypothermia persists, the infant will be transferred back to the incubator.
  Arms: Preterm infants in open coat

SUMMARY:
The goal of this randomized controlled trial without medication neither device (for procedure) is to compare the average length of hospital stay of infants weaned from the incubator at a weight greater than or equal to 1400 grams versus infants weaned at a weight greater than or equal to 1600 grams.

The main questions it aims to answer are:

* Is it possible to reduce the average hospital stay in the early weaning group compared with the standard weaning group?
* Is this procedure safe and without adverse outcomes between the two groups during the hospital stay and during the first week after discharge?

DETAILED DESCRIPTION:
Premature or low-birth-weight infants have low thermoregulatory abilities, higher risk of hypothermia and thus require a heated environment to survive. In the Neonatal Intensive Care Unit, these infants are placed from birth in an appropriately heated and humidified incubator. When they gain thermal competence they are gradually transferred to the open crib, normally when they reach a weight of about 1600-1800 grams, although the practice varies widely among neonatal units. Recent studies have concluded that clinically stable preterm infants can be transferred to an open crib at a body weight of less than 1600 grams. The abilities to maintain a normal body temperature in an open crib, good feeding autonomy, stable cardio-respiratory function, and acceptable growth rate are the physiological skills generally required for discharge of infants from the hospital.

The study compares the average length of hospital stay of infants weaned from the incubator at a weight greater than or equal to 1400 grams versus infants weaned at a weight greater than or equal to 1600 grams, as well as the incidence of adverse outcomes between the two groups (lower growth rate, inadequate breastfeeding, thermal lability and need for the incubator, readmission to the hospital) during the ward stay and during the first week after discharge, the degree of psychological stress of the parents, and the quality of the parent-child relationship in the two different groups.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weight less than 1400 grams in incubator who have reached a minimum weight of 1400 grams
* Stable clinical condition: normal heart rate and respiratory rate, No need for invasive respiratory assistance, no episodes of apnea, stable axillary temperature not less than 36.5°for at least 72 hours.
* No need for phototherapy
* Stable or increasing weight for at least 48 hours
* Signature by both parents of an informed consent

Exclusion Criteria:

* Severe congenital anomalies at birth
* Need for invasive respiratory support at the time of enrollment
* Ongoing phototherapy
* Major surgical pathology with need for surgery
* Failure by both parents to sign up for informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of average length of hospital stay of preterm infants | 72 hours after weaning from the incubator
  Compare the average length of hospital stay of infants weaned from the incubator at a weight greater than or equal to 1400 grams versus infants weaned at a weight greater than or equal to 1600 grams

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Priolo, Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS; UOC Neonatologia, Roma, Italy